CLINICAL TRIAL: NCT06578364
Title: Effect of Educational Program About Preconception Care on Knowledge and Attitude of Adolescents University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Delta University for Science and Technology (Other)
Responsible Party: Principal Investigator, Amira Hussin Hussin Mohammed, Associated professor at faculty of physical therapy, Delta University for Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Preconception Care
Record Dates: First submitted 2024-08-26; First posted 2024-08-29 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Preconception Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Educational Program about Preconception Care (Experimental)
  Interventions: Device: Educational Program about Preconception Care

INTERVENTIONS:
Device: Educational Program about Preconception Care — The educational program consisted of a single session, which included a lecture, pictures, videos, and discussions.

SUMMARY:
This quasi-experimental study used a pre-test-post-test design to assess the effectiveness of the teaching program. A sample of 400 students from El Mansoura University was selected using a simple random sample. The participants were given a pre-test questionnaire to evaluate their knowledge and attitude towards PCC. The educational program consisted of a single session, which included a lecture, pictures, videos, and discussions. The post-test was administered immediately after the program

ELIGIBILITY:
Inclusion Criteria:

* The study included males and females from the targeted colleges.
* Students from grade 1 to grade 4.
* Students who accepted to participate in the study.

Exclusion Criteria:

* Students from the medical sector.
* Students who refused to participate were excluded from the study.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
knowledge and attitude towards Preconception care (PCC) | The educational program consisted of a single session, which included a lecture, pictures, videos, and discussions. The post-test was administered immediately after the program.
  The questionnaire includes sections on socio-demographic factors, obstetrics, family planning, and disease-related factors, as well as sections for knowledge and attitude questions

CONTACTS AND LOCATIONS:
Locations (1):
- Amira Hussin Mohammed, Gamasa, Egypt

IPD SHARING:
Plan to Share IPD: No